CLINICAL TRIAL: NCT02358018
Title: 68Ga-DOTATOC for Imaging of Neuroendocrine Tumors: Expanded Access Trial
Status: No longer available | Type: Expanded Access
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-226
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neuroendocrine Tumors
Keywords: 68Ga-DOTATOC; PET/CT scan; 14-226
MeSH Terms: conditions — Neuroendocrine Tumors

INTERVENTIONS:
Drug: 68Ga-DOTATOC PET/CT Scan — Study participants will undergo the 68Ga-DOTATOC PET/CT after informed consent. The nominal injected dose will be up 3-5.5 mCi containing approximately 10 - 50 microgram of 68Ga-DOTATOC and will be injected via IV access lines. CT scans will be performed with our standard oral contrast agent (typically Omnipaque and/or barium) in accordance with our standard FDG practice unless some contraindication is present. Uptake period following injection will be 0.75-1hour. Acquisition time will be approximately ~1 hour. In patients who may not be able to lie still, anesthesia will be provided as per routine standard clinical practice.

SUMMARY:
The purpose of this study is to use a new type of scan, called 68Ga-DOTATOC PET/CT scan, instead of OctreoScan, the standard scan, to diagnose, monitor and manage your tumor. 68Ga-DOTATOC is an improved imaging agent being routinely used in many centers outside the USA, with better tumor detection than with OctreoScan.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed or suspected NET requiring 111In-pentetreotide imaging for clinical indications.
* High risk of NET because of familial predisposition with clinical findings requiring radiolabeled somatostatin imaging.
* Other somatostatin positive tumor for which 111In-pentetreotide has been used successfully (for example adult meningioma).
* Ability of subject or Legally Authorized Representative (LAR) (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Pregnant or lactating women: Pregnant women are excluded from this study because the effects of 68Ga-DOTATOC in pregnancy are not known; exceptions may be performed if expected risk outweighs the benefit. Pregnancy testing will follow MITS procedure for diagnostic reagents. Patients self report pregnancy status. If pregnant the test will not be performed unless in the clinical opinion of the attending physician the gain of the test is likely to outweigh the risk (this will be rare). If unsure whether pregnant or not then a urine or serum pregnancy will be performed.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to administration of 68Ga-DOTATOC in the mother, breastfeeding should be discontinued for at least one day if the mother receives 68Ga-DOTATOC.
* Patients that have contraindications for 111In-pentetreotide.
* Known severe allergy or hypersensitivity to oral contrast will preclude administration of such contrast (will preclude receiving oral contrast only).
* Patients with a body weight of 400 pounds or more or not able to enter the bore of the PET/CT scanner due to BMI, because of the compromise in image quality with CT, PET/CT and MRI that will result.
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Grewal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/